CLINICAL TRIAL: NCT02053194
Title: Developing Pharmacist-led Research to Educate and Sensitive Community Residents to the Inappropriate Prescription Burden in the Elderly
Brief Title: A Trial to De-prescribe Inappropriate Medications in the Community Dwelling Elderly
Acronym: D-PRESCRIBE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Cara Tannenbaum, Dr. Cara Tannenbaum, Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CIHR 201303MOP-299872-KTR
Record Dates: First submitted 2014-01-31; First posted 2014-02-03 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Inappropriate Dose of Drug Administered; Health Behavior
Keywords: Inappropriate prescribing; Health Education; Community Pharmacy Services; Medication Therapy Management; Preventive Health Services; Polypharmacy; Inappropriate prescriptions; Aged
MeSH Terms: conditions — Health Behavior; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmacist-led educational intervention (Experimental): Participants will receive an educational brochure on an inappropriate prescription they are currently taking from their pharmacists. Participants' physicians will receive an evidence-based pharmaceutical opinion for the same medication.
  Interventions: Behavioral: Pharmacist-led educational intervention
- Control (No Intervention): Participants in the control group will be wait-listed and observed for 6 months prior to receiving the intervention.

INTERVENTIONS:
Behavioral: Pharmacist-led educational intervention — 1) Educational material to participants in the form of a written educational brochure on inappropriate prescriptions that was developed and tested during the EMPOWER study. 2) Evidence-based pharmaceutical opinions sent to the treating physicians.
  Arms: Pharmacist-led educational intervention

SUMMARY:
The objective of this trial is to test the beneficial effect of a pharmacist-initiated knowledge transfer intervention to both patients and prescribers on the discontinuation of inappropriate prescriptions, compared to usual care. The investigators hypothesize that the pharmacist-led intervention will reduce inappropriate prescriptions by at least 20% over 6-months compared to usual care. The intervention consists of simultaneously educating consumers and providing physicians with an evidence-based pharmaceutical opinion on inappropriate prescriptions.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 65 years of age and older (no upper age limit)
* Individuals for whom prescription claims derive from only one pharmacy identifier
* Chronic consumption (> 3 month claims) of one of the target inappropriate prescriptions. (benzodiazepine/non benzodiazepine hypnotic, long-acting sulfonylurea oral hypoglycemic agents, anticholinergic agents (in the form of first-generation antihistamines) or Nonsteroidal anti-inflammatory drugs [NSAIDs] )
* Patients who are willing to participate in the study.

Exclusion Criteria:

* A probable diagnosis of dementia (persons without the capacity to provide informed consent), as determined by a) a prescription for memantine or a cholinesterase inhibitor; b) report from a caregiver or family-member; or c) a baseline screening score on the Folstein Mini-Mental State Exam < 24
* Inability to understand and or communicate in English and/or French
* Patients living in a long-term care facility
* Concomitant use of any antipsychotic medication

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 600 (Actual)
Dates: Start 2014-03; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Complete discontinuation of inappropriate prescriptions. | 6 months
  Provincial prescription insurance claims will be used to measure whether the inappropriate prescription has been discontinued in the intervention and control group at 6-months. Prescription data contain information on all dispensed prescriptions including drug name, dispensation date, dosage, drug form, duration and quantity of the drug dispensed, as well as the license number of the physician who wrote the prescription. Discontinuation of an inappropriate prescription will be defined as the lack of a claims renewal for that medication during a minimum of three or more consecutive months (with no subsequent renewals) during the nine months following receipt of the intervention.

SECONDARY OUTCOMES:
The frequency, timing and type of pharmaceutical opinions sent by the pharmacist to the patient's primary care physician. | 6 months
  The occurrence and delivery date of any pharmaceutical opinion sent to the patient's physician will be ascertained by the presence of a pharmacist billing claim recorded within 6 months after randomization of pharmacies to the intervention group. The type of opinion (evidence-based example provided by the research team vs customized by the pharmacist) will be ascertained by obtaining a photocopied paper copy of the pharmaceutical opinion from the patient's pharmacy record at the end of the trial (by law, the pharmacist must keep a copy in the patient's dossier). The dates of the paper copy will be matched to the date of the billing registered in the billing database to validate that the latter relates to the drug under study.
Effect of the pharmaceutical opinion on the prescriber's behaviour. | 6 months
  Pharmacists will be provided with a "study response card" to accompany any pharmaceutical opinion sent to a physician for study patients with inappropriate prescriptions. The "response card" will ask the physician to endorse one of the following three options: 1) I agree with the proposed recommendation and have signed the prescription recommendation you have provided to discontinue or substitute the inappropriate prescription 2) I will discuss with the patient at the next visit; or 3) no change required. The physician will be asked to fax back the response card to the pharmacist. A copy of all response cards received by the pharmacist will be collected by the research team at the end of the trial. The pharmacist will also be asked whether the physician acknowledged the pharmaceutical opinion in any other way. Lack of acknowledgment of the pharmaceutical opinion by the physician will be coded as a non-response.
Patient-physician encounters to discuss inappropriate prescriptions. | 6 months
  Patient visits to their primary care provider within the 6-months post-intervention will be ascertained by physician billing claims. Visits to physicians where discussions about inappropriate prescriptions occurred will be determined by patient self-report during the 6-month semi-structured telephone follow-up interview by asking whether patients met with their physician to discuss their prescriptions and what happened during these encounters. We will also query any phone call discussions with physician on this subject and conversations with pharmacists to discuss prescription changes.

OTHER OUTCOMES:
Change in risk perception around inappropriate prescriptions | Baseline, 6 months
  Baseline and post-intervention evaluation of participant's, pharmacist's and physician's beliefs about the risks associated with certain inappropriate prescriptions, as listed on the Beers Criteria of inappropriate medication in the elderly.

CONTACTS AND LOCATIONS:
Overall Officials: Cara Tannenbaum, MD, MSc, Principal Investigator — Centre de Recherche de l'Institut Universitaire de Gériatrie de Montréal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Turner JP, Martin P, Zhang YZ, Tannenbaum C. Patients beliefs and attitudes towards deprescribing: Can deprescribing success be predicted? Res Social Adm Pharm. 2020 Apr;16(4):599-604. doi: 10.1016/j.sapharm.2019.07.007. Epub 2019 Jul 10. PMID 31303479
- [Derived] Martin P, Tamblyn R, Benedetti A, Ahmed S, Tannenbaum C. Effect of a Pharmacist-Led Educational Intervention on Inappropriate Medication Prescriptions in Older Adults: The D-PRESCRIBE Randomized Clinical Trial. JAMA. 2018 Nov 13;320(18):1889-1898. doi: 10.1001/jama.2018.16131. PMID 30422193
- [Derived] Martin P, Tamblyn R, Ahmed S, Benedetti A, Tannenbaum C. A consumer-targeted, pharmacist-led, educational intervention to reduce inappropriate medication use in community older adults (D-PRESCRIBE trial): study protocol for a cluster randomized controlled trial. Trials. 2015 Jun 10;16:266. doi: 10.1186/s13063-015-0791-1. PMID 26058676